CLINICAL TRIAL: NCT07335367
Title: PRP Combined With Botulinum Toxin Type A Injection for the Treatment of Androgenetic Alopecia: A Study
Acronym: AGA
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NFEC-2025-311
Record Dates: First submitted 2026-01-05; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Androgenetic Alopecia (AGA)
Keywords: Platelet-Rich Plasma
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRP combined with Botulinum Toxin Type A treatment group (Experimental)
  Interventions: Combination Product: Injection of PRP combined with Botulinum Toxin Type A into the alopecic area(s)
- PRP-only control group (Active Comparator)
  Interventions: Other: PRP-only injection into the alopecic area

INTERVENTIONS:
Combination Product: Injection of PRP combined with Botulinum Toxin Type A into the alopecic area(s) — Treatment Protocol:
  Subjects in the PRP combined with Botulinum Toxin Type A (BTX-A) treatment group received injections using the same method and frequency as the PRP control group. For the first session, the injection consisted of 100 units of BTX-A reconstituted in 4 ml of PRP. The second and third sessions were identical to those administered to the control group (PRP injection only).
  Follow-up Assessments:
  A safety evaluation was conducted for each subject 14 days after the initial treatment, during which the investigator provided scalp care guidance. Subsequent evaluations for both safety and efficacy were performed at 1, 2, 3, and 6 months following the initial treatment.
  Arms: PRP combined with Botulinum Toxin Type A treatment group
Other: PRP-only injection into the alopecic area — Treatment Protocol for the PRP-Only Control Group:
  Subjects in the PRP-only control group will receive PRP injection therapy alone. The PRP will be administered intradermally at a depth of approximately 1.5-2.5 mm, with injection points spaced 1 cm apart, into the predefined scalp area (≥12 cm from the lateral canthus and ≥9 cm from the top of the ear, encompassing the frontal, temporal, parietal, and occipital regions). The injections will be administered at a dose of 0.1 ml/cm². The treatment regimen consists of monthly sessions, with 4 ml of PRP injected per session, for a total of 3 consecutive sessions.
  Follow-up Assessments:
  A safety evaluation will be conducted for each subject 14 days after the initial treatment, during which the investigator will provide personalized scalp care guidance. Subsequent comprehensive assessments evaluating both safety and efficacy will be performed at 1, 2, 3, and 6 months following the initial treatment.
  Arms: PRP-only control group

SUMMARY:
Research Purpose

The objective of this study is to determine the safety and efficacy of combined PRP and BTX-A injection therapy for Androgenetic Alopecia (AGA).

Study Content

This clinical trial is a randomized (1:1), multicenter, parallel-group, controlled study. AGA patients aged 18 to 60 years presenting to the participating centers will be recruited. After providing informed consent, eligible patients who meet the inclusion/exclusion criteria will be randomized in a 1:1 ratio, with separate randomization schedules for male and female patients, into either the experimental group (PRP combined with BTX-A injection) or the control group (PRP injection only). A total of 76 patients will be enrolled.

Control Group: Subjects randomized to the control group will receive PRP injection therapy. The PRP will be administered intradermally (at a depth of approximately 1.5-2.5 mm, with injection points 1 cm apart) into the scalp area (defined as ≥12 cm from the lateral canthus and ≥9 cm from the top of the ear, encompassing the frontal, temporal, parietal, and occipital regions) at a dose of 0.1 ml/cm². The treatment regimen consists of monthly injections, 4 ml per session, for a total of 3 consecutive sessions.

Experimental Group: Subjects randomized to the experimental group will receive injections using the same method and frequency as the control group. For the first session, the injection will consist of 100U of BTX-A reconstituted in 4 ml of PRP. The second and third sessions will be identical to those in the control group (PRP injection only).

Follow-up Assessments: For all subjects, a safety evaluation will be conducted 14 days after the first treatment, along with scalp care guidance provided by the investigator. Subsequent safety and efficacy assessments will be performed at 1, 2, 3, and 6 months following the initial treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who meet the diagnostic criteria for AGA, confirmed by medical history, clinical presentation, and trichoscopy, with a stage of Norwood-Hamilton III to V or Ludwig I to III.
2. Patients provide informed consent and voluntarily participate in the study.
3. A signed informed consent form is obtained.
4. Age between 18 and 60 years, in good general health.
5. No use of any medications for AGA treatment within the past 6 months.
6. Absence of alopecia areata, local infection, or neuromuscular diseases.

Exclusion Criteria:

1. Disease duration exceeding 5 years.
2. Patients who do not meet the diagnostic criteria for AGA.
3. Individuals with coagulation disorders.
4. Patients with active skin diseases or other severe systemic illnesses.
5. Patients with blood-borne infectious diseases such as Hepatitis A, Hepatitis B, HIV/AIDS, or Syphilis.
6. Use of any medications for hair loss treatment within the past 6 months.
7. Other conditions deemed by the investigator as unsuitable for participation, including but not limited to unreliable patients, or those unable to undergo or comprehend the study assessments.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 76 (Estimated)
Dates: Start 2026-01-09 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Hair density | 0 days, 14 days,1 month, 2months,3 months, 6 months
  Changes in hair density over time
hair density | 0 days, 14days,1 month, 2 months,3 months, 6 months
  Changes in hair density over time

IPD SHARING:
Plan to Share IPD: No